CLINICAL TRIAL: NCT03673852
Title: Peer Wellness Enhancement For Patients With Serious Mental Illness and High Medical Costs
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Yale University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: 2000023089; R34MH117188-01 (NIH)
Record Dates: First submitted 2018-08-09; First posted 2018-09-17 (Actual); Last update posted 2022-02-17 (Actual); Status verified 2022-02

CONDITIONS: Chronic Medical Condition
Keywords: Serious Mental Illness (SMI)

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Peer Wellness Enhancement (WE Harambee) (Other): This project employs a pragmatic, stepped wedge experimental design in which 60 BHH participants are randomly assigned to one of 3 waves of WE Harambee implementation (20 in each wave) during the 2 year study. Participants in this arm receive the WE Harambee Wellness Enhancement and are enrolled in a Behavioral Health Home. WE Harambee is a 6-month peer-delivered whole health intervention intended to address the 8 dimensions of wellness and the social determinants of health.
  Interventions: Behavioral: WE Harambee
- Behavioral Health Home enrollment (Other): In the stepped wedge experimental design, 40 participants at any time during the 2 year study are receiving only the Behavioral Health Home (BHH) intervention. The 2010 Patient Protection and Affordable Care Act (ACA) established a "health home" option under Medicaid that serves enrollees with chronic conditions including serious mental illness and chronic physical illness.
  Interventions: Behavioral: Behavioral Health Home Enrollment

INTERVENTIONS:
Behavioral: WE Harambee — WE Harambee is a 6-month intervention, comprised of twice a week group meetings for 12 weeks, followed by a second 12 weeks of individual peer coaching/navigation. WE Harambee aims to enhance access to and engagement in primary care and behavioral health services, as well as improve overall health and well-being, including the 8 dimensions of wellness and social determinants of health.
  Arms: Peer Wellness Enhancement (WE Harambee)
Behavioral: Behavioral Health Home Enrollment — A BHH is a Center for Medicaid Services program supporting Medicaid beneficiaries with complex needs, typically multiple chronic conditions impacting both physical and behavioral health. Utilizing a team-based clinical approach that includes the patient, his/her providers, and possibly family members, BHH programs target service fragmentation by linking community supports and resources as well as by enhancing the integration of primary and behavioral health care. Care Coordinators oversee and facilitate access to all services an individual needs to stay as healthy as possible, aiming to promote continuous health management not mere resolution of repeated acute episodes.
  Arms: Behavioral Health Home enrollment

SUMMARY:
This research addresses the important public health crisis that people with serious mental illness (SMI) are dying10-20 years younger than the average population, primarily due to chronic, untreated medical conditions. This proposal tests the feasibility, acceptability, engagement of target mechanisms, and preliminary effectiveness of a peer-led and peer-developed intervention to improve the health and wellness of people with SMI by addressing underlying social determinants of health. This research will provide key information about target mechanisms underlying peer interventions and establish the evidence needed to advance to a full scale clinical trial.

DETAILED DESCRIPTION:
60 Connecticut Mental Health Center patients enrolled in BHH will be recruited for the study. The research team will begin working closely with BHH data administrators and staff to start the recruitment process. A BHH data manager will create a randomly sorted list of the current BHH roster. This list will be stratified with respect to gender, race, and ethnicity so that the research team can collect a stratified sample for this research that is representative of the population. This stratified list will be given to BHH care coordinators, who will contact patients in each strata of the population and provide a brief, scripted introduction to the study, and attempt to obtain permission to contact. A flyer will be posted at the BHH program, providing information about the study for persons interested to self-refer to the research team. The research team will not have access to names of individuals on this roster, and will only be given names and contact information of individuals who provide permission to contact or who self-refer. The research team will then contact patients, provide preliminary information about the study and assessment procedures, answer any questions, and invite patients to participate. A consent and baseline interview time and date will be scheduled, at which time more detailed explanations about the study will be provided, ability to provide informed consent will be assessed, consent forms reviewed, signatures obtained, and release of information forms for retrieval of administrative data and to allow contact with BHH coordinator, if needed. BHH coordinators will continue working down the randomly sorted list to obtain permissions to contact until 60 BHH patients have enrolled and provided consent into the study. After completion of the consent process, patients will be randomly assigned into one of three waves of WE Harambee implementation and baseline interviews will be conducted. The first wave of implementation will be standard WE Harambee intervention, as implemented in our recent pilot trial (i.e., with no modifications or adaptations to design). While Wave 1 participants are receiving the group intervention (consisting of twice a week group meetings), the research team will be analyzing the administrative data and baseline interviews obtained on all 60 participants. Following completion of the 3 months, group intervention, Wave 1 participants will complete a follow-up quantitative interview and a follow-up qualitative interview to gather additional information about specific aspects of the intervention that have worked well, areas for improvement, and questions related to feasibility and acceptability of the intervention thus far. Wave 1 participants will then be offered 1:1 peer mentorship/coaching with a peer leader of his/her choice. Individual peer mentoring will be offered for the next three months. During this time, the research team and stakeholder advisory group will be analyzing the 3-month follow-up data, graphing mean changes from baseline in the targets of the intervention, and analyzing the qualitative interviews. The stakeholder advisory group members are people that have lived experience with both mental and primary healthcare problems. The stakeholder advisory group member's experience navigating the healthcare system will guide the research, providing special attention to the challenges, barriers and facilitators that stakeholders experienced in their journey of healthcare. The data will be shared with the stakeholder advisory group and, in tandem with the research team, identify initial modifications that can be made to the WE Harambee intervention, that can be instituted in Wave 2 administration. As Wave 1 participants are nearing completion of the 12-week individual peer mentoring phase, research team will contact all 60 participants to schedule Time 2 (T2) interviews. The interviews will occur after Wave 1 participants fully complete the intervention and will mirror the baseline (T1) and post-group interview. Adaptations will be formalized for the Wave 2 implementation, which will begin in month 10 of the study. The research process will proceed in a similar manner, with all Wave 2 participants completing a post-group interview and a qualitative interview. Analyses and interpretation of data collected to date will occur while Wave 2 participants are receiving the 1:1 peer mentoring component of the WE Harambee intervention. Adaptations will again be made, this time greater attention will be paid to measures of fidelity and changes to be reflected in the intervention manual, although any changes in process, assessment, or implementation that improves the fit of the intervention will also be made. All 60 participants will complete a T3 assessment following completion of Wave 2. Final adaptations will be made to intervention and tools and in month 17, the third and final wave of 20 participants will be offered the refined intervention. As before, Wave 3 participants will complete a post-group interview and qualitative interviews following completion of the group component of the intervention. Data will be analyzed and interpreted and final adjustments will be made, in conjunction with the stakeholder advisory board, to the implementation manuals, fidelity tools, assessment protocols, and recruitment strategies, in preparation for a full-scale clinical trial. A final assessment will be completed with all 60 participants following the end of Wave 3 (T4; month 23). Recruitment and timeline will be analyzed for between and within-Wave comparisons in target engagement and outcomes. If the hypothesized targets are engaged (i.e., participants demonstrate improvement in the direction expected) and if there is some evidence of the association between target engagement and outcomes, the researchers will move forward with plans to launch full-scale clinical trial. In brief, all 60 patients enrolled in the study will participate in individual interviews in 4 different time periods of the study: T1 (before Wave 1), T2 (after Wave 1 and before Wave 2), T3 (after Wave 2 and before Wave 3), and T4 (after Wave 3). Additionally, each participant will have one additional interview following completion of the group component of the WE Harambee intervention. The post-intervention interviews will be administered to all 60 participants who have completed the group intervention. Thirty Participants will also be invited to participate in a qualitative interview (n=20 from Wave 1, n=5 from Wave 2, n=5 from Wave 3) . The wave-specific interviews are designed to provide within-group, preliminary data that can be used to inform any adaptations/modifications to subsequent waves of intervention.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be CMHC enrolled patients in the Behavioral Health Homes Program over the age of 18 years old

Exclusion Criteria:

* Participants who are not CMHC enrolled patients in the Behavioral Health Homes Program and under the age of 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-12-06 (Actual); Primary Completion 2021-05-30 (Actual); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Self-reported coping and problem solving | 21 months
  Coping and problem solving will be measured by the Health Problem-Solving Scale (HPSS). The HPSS assesses effective and ineffective approaches to managing health-related problems. It has been used with diverse samples, including with samples from HIV and DM. Internal reliability coefficients were comparable in the two samples (HIV and Diabetes) and were within an acceptable psychometric range 0.63-0.88. Scale items range from 0 (not at all true for me) to 4 (extremely true of me). Higher scores indicate greater health problem solving. The total score will be represented by a mean value so the range of the total score is also 0-4.
Self-reported self-efficacy | 21 months
  Self-efficacy will be measured by the Self-Efficacy for Chronic Illness Management scale, a 6-item measure that assesses confidence in one's ability to manage \ symptoms, function emotionally and instrumentally, and communicate effectively with physicians. Internal consistency is reported to be .91. Scale items range from 1 (not at all confident) to 10 (totally confident). Higher scores indicate greater reported self-efficacy in managing one's chronic illness. The total score will be represented by a mean value so the range of the total score is also 0-10.
Self-reported hope | 21 months
  Hope will be measured by the Hope Scale, a 12-item measure that assesses a) agency (goal-directed determination) and b) pathways (planning ways to meet goals). Item ratings range from 1 (definitely false) to 8 (definitely true) with higher scores indicating more hope. Subscales and total scores will be represented by means so the range is also 1 to 8.
Self-reported social support | 21 months
  Social support will be assessed using the Interpersonal Support Evaluation List (ISEL). This 40-item instrument measures perceived availability of four types of support-tangible support, appraisal support, self-esteem support, and belonging support. Item ratings are 0 (false) or 1 (true), with higher scores indicating more social support. Subscales and total scores will be represented by means, accounting for missing data, so the range is also 0 to 1.
Self-reported sense of community | 21 months
  Sense of community will be measured by the Community Connections Index, a 15-item measure grounded in social capital and community capacity theories organized into two dimensions of community connections - Community engagement (8 items) and Sense of community (7 items). Item ratings range from 1 (never) to 4 (often), with higher scores indicating more community connection. The total score will be represented by a mean value so the range is also 0 to 4.
Self-reported empowerment | 21 months
  Empowerment will be measured the Empowerment Scale, which measures the construct of personal empowerment from the person's perspective. Internal consistency for the Empowerment scale as a whole has been reported, with Cronbach's alpha coefficients = 0.86 will be used to measure empowerment. Subscales include self-esteem/self-efficacy, power, community activism and autonomy, optimism and control over the future, and righteous anger. Item responses range from 1 (strongly disagree) to 4 (strongly agree), with higher scores indicating more empowerment. Subscales and total scores will be represented by a mean value, accounting for missing data, so their range is also 1-4.
Self-reported patient activation | 21 months
  Patient activation will be assessed via the Short Form version of the Patient Activation Measure (13 items). Cronbach's alpha = -.83. Item ratings range from 1 (strongly disagree) to 5 (strongly agree), with higher scores indicating more activation. The total score will be represented by a mean value accounting for missing data, so the range is also 1-5.
Self-reported health literacy | 21 months
  Health Literacy will be measured by the reading comprehension section of the Short-Test of Functional Health Literacy (S-TOFHLA), which was designed to measure the ability to read and understand things patients commonly encounter in the healthcare setting. The reading comprehension section asks respondents to read two passages about medical care and answer 20 questions in which they choose the correct missing word(s) from the sentences. Total scores range from 0-100, with 5 points given for each question correctly answered. Scores from 0-50 indicate inadequate health literacy, scores from 51-65 indicate marginal health literacy, and scores from 66-100 indicate adequate health literacy.
Self-reported barriers and facilitators to healthcare | 21 months
  Barriers and Facilitators of Healthcare will be assessed via the Peer Health Navigator Toolbox Barriers and Facilitators Measure. Internal consistency is estimated at .69. Scores range from 2 (major barrier) to 0 (not at all a barrier); 2 (helps a lot) to 0 (does not help), with higher scores indicating greater barrier or facilitator. Individual barriers and facilitators will be analyzed separately. Also, separate scores will be calculated for total barriers and total facilitators as mean scores, accounting for missing data, and will range from 0 to 2.

SECONDARY OUTCOMES:
Self-reported illness self management | 21 months
  Illness self-management will be assessed using the Coping and Stress Reduction subscales of the Strategies Used by People to Promote Health (SUPPH-29). The scale was designed specifically for people with chronic conditions, and has been used with cancer patients, patients with end stage renal disease, stroke survivors, and women with AIDS. The measure asks about how confident a person is in using different techniques to reduce stress and cope with their illness. Item ratings range from 1 (very little confidence) to 5 (quite a lot of confidence), with higher scores indicating more confidence. Subscale scores and total scores will be represented by mean scores, accounting for missing data, and will also range from 1 to 5.
Self-reported engagement in healthcare | 21 months
  Engagement in healthcare will be assessed via the Patient Health Engagement Measure. Items ask about how emotionally overwhelmed patients get when dealing with their illness. Item ratings range from 1 (very upset/discouraged) or 4 (very positive/optimistic) with higher scores indicating more positive feelings. Total scores will be represented by a mean score and will also range from 1 to 4.
Number of preventive care/screenings conducted | 21 months
  Number of preventive care/screenings conducted will be collected via electronic health records.
Number of outpatient visits | 21 months
  Number of outpatient visits will be collected via electronic health records.
Diastolic blood pressure level | 21 months
  Diastolic blood pressure will be measured in mmHg (millimeters of mercury) and collected from the participant's electronic medical record.
Systolic blood pressure level | 21 months
  Systolic blood pressure will be measured in mmHg (millimeters of mercury) and collected from the participant's electronic medical record.
hgA1c level | 21 months
  Glycated haemoglobin (hgA1c) levels will be measured in mmol/mol units and collected from the participant's electronic medical record.
Triglyceride level | 21 months
  Triglyceride levels will be measured in milligrams per deciliter (mg/dL) and collected from the participant's electronic medical record.
High-density lipoprotein (HDL) level | 21 months
  HDL levels will be measured in milligrams per deciliter (mg/dL) and obtained from the participant's electronic medical record.
Low-density lipoprotein (LDL) levels | 21 months
  LDL levels will be measured in milligrams per deciliter (mg/dL) and obtained from the participant's electronic medical record.
Body mass index (BMI) level | 21 months
  BMI levels will be measured in kilograms per square meter (kg/m2) and collected from the participant's electronic medical record.
Self-reported psychiatric symptoms | 21 months
  Psychiatric symptoms will be assessed through multiple subscales of the Symptom Checklist-90-Revised. We will collect subscales related to the symptoms we expect will be affected by Harambee: Anxiety, Depression, Psychoticism, Paranoia, Somatization, Hostility, Interpersonal sensitivity, and Obsessive-compulsiveness. Internal consistency of the subscales is high (range .77-.90). Item scores range from 1 (not at all) to 5 (extremely).
Self-reported substance use | 21 months
  Substance use will be assessed using the Addiction Severity Index. The ASI is a structured interview for evaluating the degree of potential treatment barriers across domains typically affected by alcohol and drug use disorders, including psychiatric and social considerations. For the purposes of this investigation, we will limit administration to the alcohol and drug use subscales. The alcohol and drug subscales concern the frequency and severity of use in the past 30 days. The ASI has been rigorously assessed within similar client populations and shown to demonstrate high reliability for assessing alcohol and drug use and its consequences, Cronbach alpha = 0.65-0.89. Item ratings range from 0 (not at all) to 4 (extremely).
Self-reported quality of functioning | 21 months
  Functional status will be assessed by the Quality of Well-being scale (QWB-SA), a common health related quality of life measuring health utilities. Most scores are coded 0 (no) or 1 (yes). Overall, the QWB-SA includes five parts assessing physical and mental health symptoms (chronic and acute), self-care, mobility, physical functioning, and social activities. In all, the domain scores are combined into a single index score ranging from 0.09 (lowest possible health state) to 1 for perfect health.
Self-reported overall wellness | 21 months
  Overall Wellness will be measured by the 8 Dimensions of Wellness Measure. This measure assesses the extent to which respondents engage in behaviors that promote physical, intellectual, environmental, spiritual, emotional, financial, social, and occupational wellness. Item ratings range from 4 (always true) to 1 (never true), with higher scores indicating greater wellness. Subscale and total scores are represented by mean scores, accounting for missing data, and have the same range of 1 to 4.
Number of Emergency Department visits | 21 months
  Number of Emergency Department visits will be collected via electronic health records.
Number of Hospitalizations | 21 months
  Number of Hospitalizations will be collected via electronic health records.

CONTACTS AND LOCATIONS:
Overall Officials: Chyrell D Bellamy, Ph.D., Principal Investigator — Yale University
Locations (1):
- CT Mental Health Center, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes
Research Resources generated will be freely distributed to qualified academic investigators for non-commercial research. Materials generated will be disseminated in accordance with University/Participating institutional and NIH policies. Depending on such policies, materials may be transferred to others under the terms of a material transfer agreement. Access to databases and associated software tools generated under the project will be available for educational, research and non-profit purposes. Such access will be provided using web-based applications, as appropriate, to avoid or minimize associated costs.
  Research data which documents, supports and validates research findings will be made available after the main findings from the final research data set have been accepted for publication. All data obtained from participants will also be shared via the NDCT related to Mental Illness. In enrolling participants, necessary information will be obtained to generate a GUID.
Supporting Information: Study Protocol, ICF
Time Frame: Data will become available at the completion of data analysis and final report indefinitely.
Access Criteria: The research generated will be freely distributed to qualified academic investigators for non-commercial research. Materials generated will be disseminated in accordance with University/Participating institutional and NIH policies. Interested parties my also contact the Principal Investigator for information.